CLINICAL TRIAL: NCT01494480
Title: The Clinical Study on the Use of Umbilical Cord Mesenchymal Stem Cells in Amyotrophic Lateral Sclerosis
Brief Title: The Clinical Trial on the Use of Umbilical Cord Mesenchymal Stem Cells in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20111207ALS
Record Dates: First submitted 2011-12-07; First posted 2011-12-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; stem cell
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell transplantation (Experimental): After stem cell prepared, the patients accepted 4 times stem cell transplantations through lumbar puncture, the time is 3-5days between two treatments. The patient would have to be in the bed at least 6 hours and removed the pillow.
  Interventions: Procedure: stem cell transplantation

INTERVENTIONS:
Procedure: stem cell transplantation — after stem cell prepared, the patients accepted 4 times stem cell transplantations through lumbar puncture, the time is 3-5days between two treatments. The patient would have to be in the bed at least 6 hours and removed the pillow.
  Other Names: the stem cell treatment of ALS

SUMMARY:
Patients with Amyotrophic Lateral Sclerosis (ALS) typically endure a progressive paralysis due to the continued loss of motoneurons that leads them to death in less than 5 years. No treatment has changed its natural history. Intrathecal injection of umbilical cord mesenchymal stem cells can secret trophic factors that keep the motorneurons functional. The investigators have designed a phase I/II clinical trial to check the feasibility of this approach in humans.

DETAILED DESCRIPTION:
A total of 30 diagnosed ALS patients. The patients would got these symptoms such as gait difficulty and tremor, hand incoordination or speech difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose established following the World Federation of Neurology criteria
* More than 6 and less than 36 months of evolution of the disease
* Medullar onset of the disease
* More than 20 and less than 65 years old
* Forced Vital Capacity equal or superior to 50%
* Total time of oxygen saturation <90% inferior to 2% of the sleeping time
* Signed informed consent

Exclusion Criteria:

* Neurological or psychiatric concomitant disease
* Need of parenteral or enteral nutrition through percutaneous endoscopic gastrostomy or nasogastric tube
* Concomitant systemic disease
* Treatment with corticosteroids, immunoglobulins or immunosuppressors during the last 12 months
* Inclusion in other clinical trials
* Unability to understand the informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Nerve functional evaluation | within one week before,1month,6months,12months and 24months after transplantation
  1. Medical Research Council scale：To determine the strength of bilateral little finger abductor muscle and anterior tibial.
  2. To evaluate the situation of upper motor neuron impairment through the Ellis reflex scale
  3. The severity evaluation: NorrisALS score and ALS functional rating scale, ALSFRS
  4. Speed of disease progression by the following formula：Progress rate = (40-ALSFRS score) / course
  5. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI) and memory (Mini Mental State Examination)
Forced vital capacity | within one week before,1month,6months,12months and 24months after transplantation
  vital capacity(VC）、forced vital capacity( FVC）、forced expiratory volune(FEV1）、FEV1/FVC、maximal voluntary ventilation(MVV）、peak expiratory flow(PEF）

SECONDARY OUTCOMES:
Blood test | within one week before,1month,6months,12months and 24months after transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers , Lymphocytes classification, cholesterol total、Triglyceride、low density lipoprotein、Glycosylated serum protein glycosylated hemoglobin、Islet function，Na+、K+
Urinal test | within one week before,1month,6months,12months and 24months after transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin. CSF test:：IgA, IgG quantitation
Electrophysiology examination | within one week before,1month,6months,12months and 24months after transplantation
  motor evoked potential(MEP)、nerve conduction and electromyologram(EMG)

CONTACTS AND LOCATIONS:
Overall Officials: YiHua An, Study Director — Chinese People's Armed Police Force
Locations (1):
- Yihua An, Beijing, China